CLINICAL TRIAL: NCT04516278
Title: A 3-month Study to Assess the Safety of ONS-5010 in Subjects With Visual Impairment Due to Retinal Disorders, NORSE THREE
Brief Title: A 3-month Study to Assess the Safety of ONS-5010 in Subjects With Visual Impairment Due to Retinal Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Outlook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONS-5010-003
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Age-related Macular Degeneration; Neovascular Age-related Macular Degeneration; Wet Macular Degeneration; BRVO - Branch Retinal Vein Occlusion; Diabetic Macular Edema
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Retinal Vein Occlusion | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Biological: bevacizumab (Experimental): ONS-5010
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — 1.25 mg, intravitreal injection
  Other Names: ONS-5010

SUMMARY:
The study will evaluate the safety of ophthalmic bevacizumab in subjects diagnosed with a retinal condition that would benefit from treatment with intravitreal injection of bevacizumab, including: exudative age-related macular degeneration, diabetic macular edema, or branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Active clinical diagnosis and OCT confirmation of one of the following retinal disorders: exudative age-related macular degeneration (AMD), diabetic macular edema (DME), or branch retinal vein occlusion (BRVO) and, in the opinion of the Investigator, requires treatment with an anti-VEGF therapy

Exclusion Criteria:

* Previous use of approved anti-VEGF or Avastin® within 4 weeks preceding randomization
* Macular edema due to something other than exudative AMD, DME or BRVO, in the study eye
* History of inadequate response to previous intravitreal anti-VEGF therapy
* History of any intraocular or periocular corticosteroid injection or implant, in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1-month preceding randomization
* Any concurrent intraocular condition in the study eye that may require medical or surgical intervention or contribute to vision loss during the study period
* Active intraocular inflammation in the study eye
* Current vitreous hemorrhage in the study eye
* Polypoidal choroidal vasculopathy (PCV) in the study eye
* History of idiopathic, infectious or autoimmune-associated uveitis in either eye
* Current ocular or periocular infection, such as conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* Current treatment for active systemic infection
* Known allergy to any component of the study drug , not amenable to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Frequency and incidence of treatment-emergent adverse events | 3 months

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Clinical Site, Tucson, Arizona
  - Clinical Site, Beverly Hills, California
  - Clinical Site, Glendale, California
  - Clinical Site, Long Beach, California
  - Clinical Site, Palm Desert, California
  - Clinical Site, Poway, California
  - Clinical Site, Clearwater, Florida
  - Clinical Site, Winter Haven, Florida
  - Clinical Site, Oak Forest, Illinois
  - Clinical Site, Springfield, Illinois
  - Clinical Site, Hagerstown, Maryland
  - Clinical Site, Albuquerque, New Mexico
  - Clinical Site, Chambersburg, Pennsylvania
  - Clinical Site, Rapid City, South Dakota
  - Clinical Site, Germantown, Tennessee
  - Clinical Site, Abilene, Texas
  - Clinical Site, Arlington, Texas
  - Clinical Site, McAllen, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Willow Park, Texas

IPD SHARING:
Plan to Share IPD: No